CLINICAL TRIAL: NCT02212054
Title: A Prospective, Randomized Controlled Trial of Conservative Versus Surgery Treatment of Children With Hirschsprung Allied Disease
Brief Title: A Trial on Treatments of Hirschsprung Allied Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Feng Jiexiong, Chief of pediatric surgery department, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101
Record Dates: First submitted 2014-08-06; First posted 2014-08-08 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Complications of Treatment; Complication of Surgical Procedure; Megacolon, Not Hirschsprung
MeSH Terms: conditions — Megacolon | interventions — Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conservative & operative treatment (Experimental): anal dilation; colon lavage; probiotics
  Interventions: Behavioral: conservative
- operative treatment (Active Comparator): one stage pull- through radical colectomy
  Interventions: Procedure: operative

INTERVENTIONS:
Behavioral: conservative — anal dilatation; colonic lavage; oral probiotic
  Arms: conservative & operative treatment
Procedure: operative — one stage pull through radical colectomy
  Arms: operative treatment

SUMMARY:
The present study was designed to compare the efficacy of conservative treatment to operative treatment for improvement of constipation symptoms in children with Hirschsprung allied disease

DETAILED DESCRIPTION:
The present study was designed to compare the efficacy of conservative treatment,such as anal dilatation, colonic lavage and so on, to operative treatment for improvement of constipation symptoms in children with Hirschsprung allied disease

ELIGIBILITY:
Inclusion Criteria:

* hard or firm stools for twice or less per week
* a predicting score of less than 5 refer to literature: Wu, X.J., et al., A new diagnostic scoring system to differentiate Hirschsprung's disease from Hirschsprung's disease-allied disorders in patients with suspected intestinal dysganglionosis. Int J Colorectal Dis, 2013. 28(5): p. 689-96

Exclusion Criteria:

* functional constipation
* a predicting score of more than 5 refer to literature: Wu, X.J., et al., A new diagnostic scoring system to differentiate Hirschsprung's disease from Hirschsprung's disease-allied disorders in patients with suspected intestinal dysganglionosis. Int J Colorectal Dis, 2013. 28(5): p. 689-96

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
the change of defecation frequency | 6~12 months
  the changes of defecation frequency at 6~12 months after treatment

SECONDARY OUTCOMES:
stool pattern | 6~12 months
  stool pattern as hard stool or loose stool
controlling stool ability | 6~12 months
  whether patients' controlling stool ability is better or not after treatment
complications | 6~12 months
  complications were suffered by patients or not

CONTACTS AND LOCATIONS:
Overall Officials: Qi T Zhu, PhD, Principal Investigator — department of pediatric surgery
Locations (1):
- Department of Pediatric Surgery, Wuhan, Hubei, China